CLINICAL TRIAL: NCT06102096
Title: A Randomized Controlled Trial of a Culturally Adapted iCBT for Arabic-speaking Refugee Youth With Common Mental Health Problems
Brief Title: Culturally Adapted iCBT for Arabic-speaking Refugee and Migrant Youth With Common Mental Health Problems
Acronym: RAHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Shervin Shahnavaz, PhD Lecturer, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KI-CNS-230918
Record Dates: First submitted 2023-10-11; First posted 2023-10-26 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-01

CONDITIONS: Depressive Symptoms; Anxiety; Insomnia; Grief; Psychological Trauma; Resilience; Stress; Marital Relationship; Psychological Well-Being
Keywords: Cognitive behavioral therapy; Psychological well-being; Resilience; Refugee; migrant; youth; mental problems
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Psychological Trauma; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Tailored iCBT for mild to moderate common mental health problems over a period ranging from 6 to 10 weeks.
  Interventions: Behavioral: Culturally Adapted iCBT
- Waiting-list (No Intervention): control group

INTERVENTIONS:
Behavioral: Culturally Adapted iCBT — A culturally adapted iCBT targeting mild to moderate mental health problems among Arabic-speaking refugee and migrant youth.
  Arms: Active group

SUMMARY:
The aim of the current study is to explore whether culturally adapted internet-based cognitive behavioral therapy is effective in reducing the symptoms of various common mental health problems among Arabic-speaking refugee and migrant youth. We hypothesize that the symptoms of the psychological problems will significantly be reduced among youth who will receive iCBT compared to youth in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 15 and 29.
* A score above the cut-off 1.75 on HSCL-25
* Has a refugee or migrant background
* Has a good and stable internet connection
* Has access to a computer, a tablet or a smartphone
* Is fluent in reading and writing Arabic
* Has the ability to dedicate time to take part in the intervention for 6-10 weeks.

Exclusion Criteria:

* Is suffering from a severe mental illness, such as psychosis or severe depression.
* Is suffering from substance abuse
* Is undergoing a psychological treatment
* Has a high risk of suicide

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
HSCL-25 | Pre-intervention, during the intervention, immediately after the intervention, 6 months after completion of the intervention
  Assessment of anxiety and depressive symptoms

SECONDARY OUTCOMES:
PHQ-9 | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  assessment of depressive symptoms
PSYCHLOPS | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Impact of problematic area on function
ISI | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Assessment of severity of insomnia
PG-13 | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Assessment of prolonged grief disorder
PCL-5 | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  assessment of symptoms of post-traumatic stress disorder
WHO-5 | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  assessment of subjective psychological well-being
BRS | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  assessment of resilience

OTHER OUTCOMES:
CSQ | immediately after the intervention, 6 months after completion of the intervention
  assessment of the levels of satisfaction of the participant with the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Demetry Y, Wasteson E, Lindegaard T, Abuleil A, Geranmayeh A, Andersson G, Shahnavaz S. Individually Tailored and Culturally Adapted Internet-Based Cognitive Behavioral Therapy for Arabic-Speaking Youths With Mental Health Problems in Sweden: Qualitative Feasibility Study. JMIR Form Res. 2023 Nov 24;7:e46253. doi: 10.2196/46253. PMID 37999955
- [Background] Lindegaard T, Wasteson E, Demetry Y, Andersson G, Richards D, Shahnavaz S. Investigating the potential of a novel internet-based cognitive behavioural intervention for Dari and Farsi speaking refugee youth: A feasibility study. Internet Interv. 2022 Apr 1;28:100533. doi: 10.1016/j.invent.2022.100533. eCollection 2022 Apr. PMID 35433279
- See also: Registration page — http://rahaarabi.com
- See also: About the research project — https://liu.se/en/research/saha